CLINICAL TRIAL: NCT07176299
Title: Efficacy of Unilateral Laparoscopic Transversus Abdominis Plane Block Compared to Local Infiltration in Postoperative Analgesia Following Laparoscopic Cholecystectomy
Brief Title: Unilateral Laparoscopic TAP Block vs. Local Infiltration in Post-Cholecystectomy Analgesia
Acronym: TAP vs LAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warmia and Mazury in Olsztyn (Other)
Responsible Party: Principal Investigator, Łukasz Dyśko, Principal Investigator, University of Warmia and Mazury in Olsztyn
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: University of Warmia and Mazur
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cholelithiasis; Cholecystectomy, Laparoscopic; Pain, Postoperative; Anesthesia, Local; Nerve Block
Keywords: Laparoscopic cholecystectomy; unilateral transversus abdominis plane block; local anesthetic infiltration; postoperative pain management; regional anesthesia
MeSH Terms: conditions — Cholelithiasis; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a 1:1:1:1 ratio to one of four parallel groups:
  1. unilateral laparoscopic TAP block,
  2. local anesthetic infiltration (LAI),
  3. combined TAP+LAI,
  4. control (no regional anesthesia).
  Each participant remained in the assigned group throughout the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients were blinded to group allocation. The statistician analyzing the results was also blinded. Care providers performing the procedures were not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- TAP Block (Experimental): Participants received a unilateral laparoscopic transversus abdominis plane (TAP) block performed under direct laparoscopic vision using 20 mL of 0.25% bupivacaine.
  Interventions: Procedure: Unilateral laparoscopic TAP block (0.25% bupivacaine)
- Local Anesthetic Infiltration (LAI) (Active Comparator): Participants received local infiltration of 20 mL of 0.25% bupivacaine at the trocar insertion sites under laparoscopic guidance.
  Interventions: Procedure: Local anesthetic infiltration (0.25% bupivacaine)
- TAP + LAI (Experimental): Participants received a combination of unilateral laparoscopic TAP block (10 mL of 0.25% bupivacaine) and local anesthetic infiltration at trocar sites (10 mL of 0.25% bupivacaine).
  Interventions: Procedure: Combined TAP block and local anesthetic infiltration (0.25% bupivacaine)
- Control (No Regional Anesthesia) (No Intervention): Participants did not receive regional anesthesia. Postoperative pain management was provided only with standardized intravenous analgesics.

INTERVENTIONS:
Procedure: Unilateral laparoscopic TAP block (0.25% bupivacaine) — Injection of 20 mL 0.25% bupivacaine into the transversus abdominis plane under direct laparoscopic vision.
  Arms: TAP Block
Procedure: Local anesthetic infiltration (0.25% bupivacaine) — Injection of 20 mL 0.25% bupivacaine distributed across trocar insertion sites under laparoscopic guidance.
  Arms: Local Anesthetic Infiltration (LAI)
Procedure: Combined TAP block and local anesthetic infiltration (0.25% bupivacaine) — 10 mL of 0.25% bupivacaine given as a TAP block and 10 mL administered as local infiltration at trocar sites.
  Arms: TAP + LAI

SUMMARY:
This study compared different methods of pain control after laparoscopic gallbladder removal. A total of 160 patients were randomly assigned to receive either a unilateral laparoscopic TAP block, local anesthetic infiltration, a combination of both, or no regional anesthesia. Pain scores, use of pain medication, and complications were measured up to 24 hours after surgery. The TAP block group experienced less pain and fewer wound-related problems, showing that this method is safe and effective for postoperative pain relief.

DETAILED DESCRIPTION:
Gallbladder stones are a common condition, and laparoscopic cholecystectomy is the standard treatment. Effective pain control after surgery is important for recovery and patient comfort. Traditionally, local anesthetic infiltration (LAI) at the surgical wound sites is used. Another method, the transversus abdominis plane (TAP) block, may provide better pain relief.

This prospective, randomized clinical trial was conducted at the University Clinical Hospital in Olsztyn, Poland. A total of 160 patients undergoing elective laparoscopic cholecystectomy were randomized into four groups: TAP block, LAI, TAP+LAI, and control. All patients received the same type of anesthesia and standard pain medications.

The primary goal was to compare pain intensity within 24 hours after surgery using the Numerical Rating Scale (NRS). Secondary measures included use of additional painkillers, recovery scores (Aldrete), and possible complications at the wound site. The influence of surgical drains and gallstone size on pain was also examined.

The study found that the unilateral laparoscopic TAP block provided the best pain relief, fewer wound-related complications, and reduced need for additional medications compared with other methods. These results suggest that the laparoscopic TAP block is a safe and effective option for improving postoperative pain management after gallbladder surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 to 85 years
* Scheduled for elective laparoscopic cholecystectomy for symptomatic cholelithiasis confirmed by ultrasonography
* American Society of Anesthesiologists (ASA) physical status I-II
* Provided written informed consent

Exclusion Criteria:

* ASA physical status III-IV
* Contraindications to laparoscopy
* Acute cholecystitis diagnosed preoperatively or perioperatively
* Chronic analgesic use
* Spinal degenerative joint disease
* Known allergy to local anesthetics
* Opioid or alcohol dependence
* Psychiatric or neurological disorders
* Lack of consent or withdrawal of consent

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity measured by Numerical Rating Scale (NRS) at 2, 6, and 24 hours after laparoscopic cholecystectomy | Pain scores were recorded at 2 hours, 6 hours, and 24 hours after laparoscopic cholecystectomy during the first postoperative day.
  Pain intensity was assessed using the Numerical Rating Scale (NRS), where 0 = no pain and 10 = worst imaginable pain. Scores were recorded by patients at rest at three time points after laparoscopic cholecystectomy: 2 hours, 6 hours, and 24 hours postoperatively. Pain was evaluated as an overall score and at specific surgical sites (umbilical, subcostal, and substernal wounds). Assessments were performed only when patients reached an adequate level of consciousness, verified by Aldrete score.

SECONDARY OUTCOMES:
Use of rescue analgesics (metamizole, paracetamol, oxycodone) within 24 hours after laparoscopic cholecystectomy | Rescue analgesic use assessed at 6, 12, 18, and 24 hours after surgery during the first postoperative day.
  Rescue analgesic use was recorded for each participant during the first 24 hours after laparoscopic cholecystectomy. Medications included metamizole, paracetamol, and oxycodone, administered according to standardized postoperative pain protocols: metamizole at 6, 12, 18, and 24 hours unless NRS ≤1, paracetamol if NRS >4, and oxycodone if NRS >6. The number and percentage of patients requiring each medication at 6, 12, 18, and 24 hours postoperatively were analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Hospital in Olsztyn, Olsztyn, Warmian-Masurian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this was a single-center clinical study and data contain sensitive patient information that cannot be fully anonymized for public release.